CLINICAL TRIAL: NCT05420298
Title: Short Term Effect of Cervical Mobilization vs Manipulation on Blood Pressure in Hypertensive Subjects( Randomized Control Trial)
Brief Title: Short Term Effect of Cervical Mobilization vs Manipulation on Blood Pressure in Hypertensive Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed El-Moatasem Mohamed, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003253
Record Dates: First submitted 2022-06-08; First posted 2022-06-15 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical mobilization (Experimental): session will include3-5 repetitions of muscle energy technique in combination of facet joint mobilization of unilateral antro-posterior glide and extension repetitions
  Interventions: Other: cervical mobilization
- cervical manipulation (Active Comparator): patients will receive high velocity low amplitude thrust
  Interventions: Other: cervical manipulation

INTERVENTIONS:
Other: cervical mobilization — All participants will receive only single session of cervical mobilization
  Arms: cervical mobilization
Other: cervical manipulation — All participants will receive only single session of cervical manipulation
  Arms: cervical manipulation

SUMMARY:
Spinal pain or misalignment is a very common disorder affecting a significant number of populations resulting in substantial disability and economic burden. Various manual therapeutic techniques such as spinal manipulations and mobilizations can be used to treat and manage pain and movement dysfunctions such as spinal malalignments and associated complications. These manual therapeutic techniques can affect the cardiovascular parameters .

-

DETAILED DESCRIPTION:
Group A group (n=20). All participants will receive only single session of neck mobilization. Grade IV unilateral posteroanterior pressure and sustained extension to be applied restricted joints and muscle energy technique.

- Group B (n=20) will receive single session of neck manipulation with high-velocity, low-amplitude thrust over restricted joints (one at a time) with the goal of restoring normal range of motion in the joint.

ELIGIBILITY:
Inclusion Criteria:

* SBP ranging from 135 to 159 mm Hg or DBP ranging from 85 to 99 mm Hg over 3 qualifying BP screening visits
* The age of participants will range from 27 to 60 years old.
* Body mass index of participants will range between < 39 kg/m².

Exclusion Criteria:

* cardiovascular diseases or surgery, including second- or third-degree heart block, angina pectoris, defibrillator, valvular disease, recent myocardial infarction, cardiac surgery in the past 12 months.
* history of stroke.
* body mass index (BMI) greater than 39 kg/m2.
* pregnancy.

Ages: 27 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure measurement | it will be measured immediately before and after single session treatment
  systolic pressure - the pressure when your heart pushes blood out and is measured by Mercury sphygmomanometer and stethoscope

SECONDARY OUTCOMES:
diastolic blood pressure | it will be measured immediately before and after single session treatment
  the pressure when your heart rests between beats is measured by Mercury sphygmomanometer and stethoscope
oxygen saturation | it will be measured immediately before and after single session treatment
  Oxygen saturation is a vital parameter to define blood oxygen content and oxygen delivery and is measured by pulse oximetry
perfusion index | it will be measured immediately before and after single session treatment
  Perfusion index is an indication of the pulse strength at the sensor site. The PI's values range from 0.02% for very weak pulse to 20% for extremely strong pulse.Perfusion index is normally monitored with pulse oximeters
pain assessment | it will be measured immediately before and after single session treatment
  The visual analog scale (VAS) is a tool widely used to measure pain

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt